CLINICAL TRIAL: NCT00724646
Title: Direct Care Staff and Parents'/Legal Guardians' Perspectives on End-of-Life Care in a Long-Term Care Facility for Medically Fragile and Intellectually Disabled Pediatric and Young Adult Residents
Brief Title: Perspectives on End-of-Life Care for Medically-Fragile Children and Young Adults
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Richard Grossberg, MD, Hattie Larlham Center for Disabled Children
Other Study IDs: End-of-Life Care
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Death
Keywords: parents; medically fragile; death; end-of-life care; surveys
MeSH Terms: conditions — Death | interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Habilitation assistants
  Interventions: Other: Survey; Other: Focus group
- 2: Parents/ legal guardians
  Interventions: Other: Survey; Other: Focus group

INTERVENTIONS:
Other: Survey — 3 individual surveys
Other: Focus group — Focus group discussions facilitated by a psychologist

SUMMARY:
Hattie Larlham is a specialized long-term care facility for pediatric and young adult residents who are medically fragile and intellectually disabled, whose daily care is provided by direct care staff, Habilitation Assistants (HA), in conjunction with nurses and other direct care providers. The purpose of this study is to assess the perspectives of HA and parents/legal guardians on end-of-life care in a long-term care facility for pediatric and young adult residents who are medically fragile and intellectually disabled.

ELIGIBILITY:
Inclusion Criteria:

* HA at Hattie Larlham between January 1, 2006 to present
* HA provided care to > 1 resident whose death occurred between January 1, 2006 through the end of the study period
* HA provided ongoing care to the resident for at least 5 days in the last 30 days at Hattie Larlham before the resident's death
* Parent/legal guardian of a Hattie Larlham resident whose death occurred between January 1, 2006 through the end of the study

Exclusion Criteria:

* HA employed < 30 days at Hattie Larlham or cared for resident <5 days in last 30 days prior to the resident's death
* HA or parent/legal guardian who has not experienced a Hattie Larlham resident's death since December 31, 2005

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents/ legal guardians and habilitation assistants
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Participants' responses to survey questions. | Start of Study

SECONDARY OUTCOMES:
Participants' responses to focus group discussions. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Richard Grossberg, MD, Principal Investigator — Hattie Larlham Center for Disabled Children
Locations (1):
- Hattie Larlham Center for Disabled Children, Mantua, Ohio, United States

REFERENCES:
- [Background] Brazil K, McAiney C, Caron-O'Brien M, Kelley ML, O'Krafka P, Sturdy-Smith C. Quality end-of-life care in long-term care facilities: service providers' perspective. J Palliat Care. 2004 Summer;20(2):85-92. PMID 15332472
- [Background] Contro N, Larson J, Scofield S, Sourkes B, Cohen H. Family perspectives on the quality of pediatric palliative care. Arch Pediatr Adolesc Med. 2002 Jan;156(1):14-9. doi: 10.1001/archpedi.156.1.14. PMID 11772185
- [Background] Vohra JU, Brazil K, Szala-Meneok K. The last word: family members' descriptions of end-of-life care in long-term care facilities. J Palliat Care. 2006 Spring;22(1):33-9. PMID 16689413